CLINICAL TRIAL: NCT04943380
Title: An Observational Study of Efficacy and Utility of Cxbladder Tests in the Identification of Low vs High Risk Patients and the Detection of Urothelial Carcinoma in Patients Presenting With Hematuria
Brief Title: Efficacy and Utility of Cxbladder Tests in Hematuria Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CXB/2019/VA
Record Dates: First submitted 2020-03-02; First posted 2021-06-29 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hematuria; Urothelial Carcinoma
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A minimum of 30 mL of urine will be required for the sampling system to function. Two 5 mL aliquots of the collected urine will be transferred to a vacutainer containing a preservative reagent, and couriered to Pacific Edge Diagnostic NZ Laboratories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hematuria undergoing investigation for UC: Patients will be recruited from those presenting with hematuria and undergoing investigative cystoscopy for the determination of possible urothelial carcinoma. This includes patients referred via imaging or from other departments for assessment of hematuria. Microscopic hematuria is defined as > 3 red blood cells per high-powered microscopy field for a properly collected urine sample.
  Interventions: Diagnostic Test: Cxbladder

INTERVENTIONS:
Diagnostic Test: Cxbladder — The Cxbladder Detect test, developed by Pacific Edge Ltd (O'Sullivan 2012; Holyoake 2008; National Health Committee 2015b) is a molecular diagnostic test, which consists of five mRNA transcripts measured in a small volume of urine.

SUMMARY:
Prospective observational study to validate the performance characteristics and clinical utility of Cxbladder tests in a Veterans Affairs cohort.

DETAILED DESCRIPTION:
Non-invasive, voided urine sample used for both Cxbladder molecular tests, voided urine sample may be used for standard of care testing. Retrospective analysis of data after study completion ensures a de-phasing of study sample analysis from clinical decision making; patient treatment and management.

The study aims to sequentially recruit up to 1000 patients presenting for assessment of hematuria (microscopic or macroscopic) by cystoscopy across multiple Veterans Affairs sites

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing investigation of recent confirmed hematuria (by either flexible or rigid cystoscopy/TURBT), including hematuria patients referred due to suspicious/positive imaging, in order to determine the presence of urothelial carcinoma.
* Able to provide a voided urine sample of the required minimum volume
* Able to give written consent
* Able and willing to comply with study requirements
* Aged 18 years or older

Exclusion Criteria:

* Prior history of bladder malignancy, prostate or renal cell carcinoma
* Prior genitourinary manipulation (flexible or rigid cystoscopy / catheterisation, urethral dilation) in the 14 days before urine collection
* Previous alkylating based chemotherapy
* Known Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted with all hematuria patients who present to an outpatient clinic to undergo clinical assessment including cystoscopy and who fulfil study requirements. Consented eligible patients will attend their scheduled clinic visit and undergo all standard tests as clinically indicated.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with bladder cancer who are correctly identified as having cancer (true positives) and no cancer (true negatives) by the Cxbladder test. | The outcome measure will be assessed by 6 months after trial completion.
  The Cxbladder test results will be compared to that of cystoscopy, which is the gold standard method for diagnosing urothelial cancer; the true positive and true negative rates will be measured, along with the false positive and false negative rates of the test. The results will be reported as sensitivity and specificity of the Cxbladder test for detecting urothelial cancer in patients with hematuria
Probability that patients identified as having cancer and no cancer by the Cxbladder test truly have cancer (positive predictive value; PPV), and truly have no cancer (negative predictive value; NPV) respectively. | Time Frame: The outcome measure will be assessed by 6 months after trial completion.
  The Cxbladder test results will be compared to that of cystoscopy, which is the gold standard method for diagnosing urothelial cancer; the true positive and true negative rates will be measured, along with the false positive and false negative rates of the test. The results will be reported as sensitivity and specificity of the Cxbladder test for detecting urothelial cancer in patients with recurrent disease.

SECONDARY OUTCOMES:
Comparison of the Cxbladder test's sensitivity, specificity, PPV and NPV with that of Cytology. | The outcome measure will be assessed by 6 months after trial completion.
  Performance characteristics (sensitivity, specificity, PPV and NPV) of the Cxbladder test for detecting recurring urothelial cancer will be compared to urine cytology, in addition to the gold standard test (cystoscopy). All comparator tests will be carried out on the same voided urine sample used for Cxbladder tests.
To compare the theoretical clinical outcome of patients tested using Cxbladder tests | The outcome measure will be assessed by 6 months after trial completion.
  To compare the theoretical clinical outcome of patients tested using Cxbladder tests in combination (Triage followed by Detect and / or Resolve) before investigative cystoscopy with evaluation by (positive, negative or suspicious) cystoscopy alone to establish the true proportion requiring cystoscopy, thereby determining the potential of Cxbladder to reduce or adjudicate the cystoscopy burden of hematuria patients and/or sub cohorts under clinical evaluation in a hospital urology clinic setting.
To compare the theoretical clinical outcome of patients tested using Cxbladder signatures before investigative cystoscopy with evaluation by cystoscopy alone to establish the true proportion requiring cystoscopy. | The outcome measure will be assessed by 6 months after trial completion.
  To compare the theoretical clinical outcome of patients tested using Cxbladder signatures before investigative cystoscopy with evaluation by (positive, negative or suspicious) cystoscopy alone to establish the true proportion requiring cystoscopy, thereby determining the potential of Cxbladder to reduce or adjudicate the cystoscopy burden of hematuria patients and/or sub cohorts under clinical evaluation in a hospital urology clinic setting.
Performance characteristics of Cxbladder Triage and Cxbladder Detect compared with results generated at other clinical sites | The outcome measure will be assessed by 6 months after trial completion.
  To evaluate the performance characteristics of Cxbladder Triage and Cxbladder Detect compared with results generated at other clinical sites, and to the results of the pulished clinical studies by O'Sullivan et al in 2012 and Kavalieris et al in 2015

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lough, PhD, Study Chair — Pacific Edge Pty Ltd
Locations (10):
- United States (10):
  - Veterans Medical Research Foundation, San Diego, California
  - Bay Pines Veterans Affairs, Bay Pines, Florida
  - South Florida Veterans Affairs, Miami, Florida
  - James A Haley Veterans' Hospital, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - NWIHCS-Omaha VA Medical Center, Omaha, Nebraska
  - James J. Peters VAMC, New York, New York
  - Oklahoma City VA Hospital, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - White River Junction VAMC, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No